CLINICAL TRIAL: NCT01886963
Title: A Randomized, Prospective, Double-Blind Clinical Trial Using Spy Elite System in Planning Tissue Advancement Flaps and Reducing Wound Complications After Complex Ventral Hernia Repairs
Brief Title: A Clinical Trial Using Spy Elite System in Planning Tissue Advancement Flaps After Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101106A
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2021-11

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control - Blinded use of SPY Elite (Active Comparator): Group A will consist of intraoperative abdominal wall imaging prior to incision, followed by ventral hernia repair with subcutaneous advancement flaps without viewing the imaging contained within the Spy Elite system. A digital photograph will be taken before and immediately after initial incision, as well as immediately prior to and after closure. The patient will have digital photographs of the surgical wound taken by the surgical team daily until discharge, and on follow-up visits at one week, two weeks, four weeks and twelve weeks. After twenty patients have completed phase I, the surgical team will be unblinded to Spy Elite imaging. The Spy Elite imaging and all digital photographs of all patients will be reviewed.
  Interventions: Device: Control - Blinded use of SPY Elite
- SPY - Unblinded Use of SPY Elite (Experimental): Group B will have incision and advancement flap performed based on assessment of blood supply using the Spy Elite system, as well as potential flap revision if portions of the flap appear under-perfused in the pre-closure imaging. Patients will be blinded to whether or not their intraoperative Spy Elite imaging was used for operative planning. All patients will have digital photographs of the surgical wound taken by a blinded member of the surgical team daily until discharge, and on follow-up visits at one to two weeks, four weeks, and 12 weeks post-operatively. Digital photographs will be reviewed by a blinded surgeon, who will assess the wound for complications.
  Interventions: Device: SPY - Unblinded use of SPY Elite

INTERVENTIONS:
Device: SPY - Unblinded use of SPY Elite — Surgeon plans tissue advancement flaps with the aid of Spy Elite System imaging
  Arms: SPY - Unblinded Use of SPY Elite
Device: Control - Blinded use of SPY Elite — Surgeon is blinded to Spy Elite imaging and plans tissue advancement flaps according to clinical judgment alone
  Arms: Control - Blinded use of SPY Elite

SUMMARY:
The purpose of this project is to assess the efficacy of the Spy Elite System (LifeCell Corporation, Branchburg, NJ, USA) in planning tissue advancement flaps and reducing wound complications after complex ventral hernia repairs. Complex ventral hernia repairs are associated with a high rate of wound complications. To a large degree these complications are caused by creating tissue advancement flaps to close the abdomen, which can compromise the blood supply to the skin and subcutaneous tissues. The current standard of care for assessment of blood perfusion to the flaps is a surgeon's clinical judgment. It is, however, often inaccurate. The Spy Elite System was developed to address this problem. The Spy Elite System is a device that enables surgeons to visualize and evaluate tissue perfusion in real time. It can help the surgeon to identify optimal flap design and reduce the risk of postoperative wound complications related to tissue ischemia. The primary goal of this study is to evaluate the efficacy of Spy Elite System to aid a surgeon in creating tissue flaps with adequate blood supply through a prospective, randomized clinical trial. The Spy Elite System has been used successfully for assessing the viability of mastectomy flaps in breast surgery and has been shown to be extremely sensitive in predicting mastectomy flap necrosis. However, no clinical trial has been conducted in order to evaluate the efficacy of the Spy Elite System for assessing the viability of abdominal subcutaneous flaps in complex ventral hernia repairs.

DETAILED DESCRIPTION:
More than 90,000 ventral hernia repairs are performed in the US annually. Large ventral hernias often require a complex abdominal wall reconstruction including creating tissue advancement flaps. Complex abdominal wall reconstructions are associated with up to 20% rate of wound complications including skin flap necrosis and wound breakdowns. Prevention of skin necrosis and ischemia would significantly reduce the morbidity associated with these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ventral hernia that will require tissue advancement flaps at time of hernia repair
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* ASA score IV or above
* Age < 18 years
* Patients with iodine allergy
* Patients with current wound or mesh infection
* Pregnant patients
* Patients with End Stage Renal Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2011-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant T Heniford, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health - Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- SPY - Unblinded Use of SPY Elite: SPY - Unblinded use of SPY Elite will have incision and advancement flap performed based on assessment of blood supply using the Spy Elite system, as well as potential flap revision if portions of the flap appear under-perfused in the pre-closure imaging. Patients will be blinded to if intraoperative Spy Elite imaging was used. Digital photographs of the surgical wound taken by surgical team daily until discharge, and on follow-up visits post-operatively. Digital photographs will be reviewed by a blinded surgeon, who will assess the wound for complications (breakdown, necrosis, erythema, infection, or dehiscence with location specified) and assessment of healing. Upon study completion, groups will be compared for wound complications, presence of flap necrosis, quantification of flap necrosis, and healing speed.
  SPY - Unblinded Use of Spy Elite: Surgeon plans tissue advancement flaps with the aid of Spy Elite System imaging
- Control - Blinded Use of SPY Elite: Control - Blinded use of SPY Elite will consist of intraoperative abdominal wall imaging prior to incision, followed by ventral hernia repair with subcutaneous advancement flaps without viewing the imaging contained within the Spy Elite system. A digital photograph will be taken before and immediately after initial incision, as well as immediately prior to and after closure. The patient will have digital photographs of the surgical wound taken by the surgical team daily until discharge, and on follow-up visits at one week, two weeks, four weeks and twelve weeks. After twenty patients have completed phase I, the surgical team will be unblinded to Spy Elite imaging. The Spy Elite imaging and all digital photographs of all patients will be reviewed.
  Control - Blinded Use of Spy Elite: Surgeon is blinded to Spy Elite imaging and plans tissue advancement flaps according to clinical judgment alone
Period: Overall Study
Arm/Group | SPY - Unblinded Use of SPY Elite | Control - Blinded Use of SPY Elite
Started | 57 | 58
2 Week Follow Up | 55 | 55
4 Week Follow Up | 50 | 51
12 Week Follow Up | 46 | 49
Completed | 46 | 49
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Control - Blinded Use of SPY Elite: Group A will consist of intraoperative abdominal wall imaging prior to incision, followed by ventral hernia repair with subcutaneous advancement flaps without viewing the imaging contained within the Spy Elite system. A digital photograph will be taken before and immediately after initial incision, as well as immediately prior to and after closure. The patient will have digital photographs of the surgical wound taken by the surgical team daily until discharge, and on follow-up visits at one week, two weeks, four weeks and twelve weeks. After twenty patients have completed phase I, the surgical team will be unblinded to Spy Elite imaging. The Spy Elite imaging and all digital photographs of all patients will be reviewed.
  Ventral Hernia Repair with Advancement Flaps with Blinded Use of Spy Elite (Control): Surgeon is blinded to Spy Elite imaging and plans tissue advancement flaps according to clinical judgment alone
- SPY - Unblinded Use of SPY Elite: Group B will have incision and advancement flap performed based on assessment of blood supply using the Spy Elite system, as well as potential flap revision if portions of the flap appear under-perfused in the pre-closure imaging. Patients will be blinded to if intraoperative Spy Elite imaging was used. Digital photographs of the surgical wound taken by surgical team daily until discharge, and on follow-up visits post-operatively. Digital photographs will be reviewed by a blinded surgeon, who will assess the wound for complications (breakdown, necrosis, erythema, infection, or dehiscence with location specified) and assessment of healing. Upon study completion, groups will be compared for wound complications, presence of flap necrosis, quantification of flap necrosis, and healing speed.
  VHR with Advancement Flaps with Unblinded Use of Spy Elite (Experimental): Surgeon plans tissue advancement flaps with the aid of Spy Elite System imaging
- Total: Total of all reporting groups
Arm/Group | Control - Blinded Use of SPY Elite | SPY - Unblinded Use of SPY Elite | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 36 | 73
  >=65 years | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.76) | 56.7 (11.16) | 57.6 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 49 | 46 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Complications
Description: breakdown, necrosis, erythema, infection, or dehiscence with location specified
Time Frame: 12 Weeks
Measure: Number; unit: participants
Groups:
- Group A: Group A will consist of intraoperative abdominal wall imaging prior to incision, followed by ventral hernia repair with subcutaneous advancement flaps without viewing the imaging contained within the Spy Elite system. A digital photograph will be taken before and immediately after initial incision, as well as immediately prior to and after closure. The patient will have digital photographs of the surgical wound taken by the surgical team daily until discharge, and on follow-up visits at one week, two weeks, four weeks and twelve weeks. After twenty patients have completed phase I, the surgical team will be unblinded to Spy Elite imaging. The Spy Elite imaging and all digital photographs of all patients will be reviewed.
  Ventral Hernia Repair with Advancement Flaps with Blinded Use of Spy Elite (Control): Surgeon is blinded to Spy Elite imaging and plans tissue advancement flaps according to clinical judgment alone
- Group B: Group B will have incision and advancement flap performed based on assessment of blood supply using the Spy Elite system, as well as potential flap revision if portions of the flap appear under-perfused in the pre-closure imaging. Patients will be blinded to if intraoperative Spy Elite imaging was used. Digital photographs of the surgical wound taken by surgical team daily until discharge, and on follow-up visits post-operatively. Digital photographs will be reviewed by a blinded surgeon, who will assess the wound for complications (breakdown, necrosis, erythema, infection, or dehiscence with location specified) and assessment of healing. Upon study completion, groups will be compared for wound complications, presence of flap necrosis, quantification of flap necrosis, and healing speed.
  VHR with Advancement Flaps with Unblinded Use of Spy Elite (Experimental): Surgeon plans tissue advancement flaps with the aid of Spy Elite System imaging
Arm/Group | Group A | Group B
Number analyzed (Participants) | 49 | 46
participants | 16 | 17

ADVERSE EVENTS:
Time Frame: All patients had a minimum of 30 days follow up to collect for adverse events; however the mean follow up was 8.3 months for patients included in the trial analysis.
Groups:
- Control - Blinded Use of SPY Elite: Control - Blinded use of SPY Elite will consist of intraoperative abdominal wall imaging prior to incision, followed by ventra l hernia repair with subcutaneous advancement flaps without viewing the imaging contained within the Spy Elite system. A digital photograph will be taken before and immediately after initial incision, as well as immediately prior to and after closure. The patient will have digital photographs of the surgical wound taken by the surgical team daily until discharge, and on follow-up visits at one week, two weeks, four weeks and twelve weeks. After twenty patients have completed phase I, the surgical team will be unblinded to Spy Elite imaging. The Spy Elite imaging and all digital photographs of all patients will be reviewed.
  Control - Blinded Use of Spy Elite: Surgeon is blinded to Spy Elite imaging and plans tissue advancement flaps according to clinical judgment alone
Arm/Group | SPY - Unblinded Use of SPY Elite | Control - Blinded Use of SPY Elite
Serious Adverse Events (participants affected / at risk) | 5/46 | 2/49
Other Adverse Events (participants affected / at risk) | 0/46 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPY - Unblinded Use of SPY Elite (N=46) | Control - Blinded Use of SPY Elite (N=49)
Acute Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Deceased (General disorders) | 1 | 0
Vital Signs (Surgical and medical procedures) | 1 | 0 — Surgery was aborted due to abnormal vital signs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT01886963/Prot_SAP_001.pdf